CLINICAL TRIAL: NCT00460707
Title: A Phase I, Randomized, Double-Blind Study to Assess the Effects of Repeat Oral Dosing of Ketoconazole on the Pharmacokinetics of Repeat Oral Dosing of Casopitant in Healthy Subjects
Brief Title: A Study to Assess the Safety and Interaction Between Casopitant and Ketoconazole When Taken By Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: NKV109990
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: GW679769; healthy adult subjects; casopitant; ketoconazole
MeSH Terms: conditions — Nausea; Vomiting | interventions — casopitant; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): All subjects in Cohort 1 will receive ketoconazole 400 milligrams (mg) once daily on Day 1 to 9 and oral casopitant 150 mg on Day 4 and 50 mg on Day 5 and Day 6 of treatment period 1. After a washout period of 21 days, subjects will be administered oral casopitant 150 mg on Day 1 and 50 mg on Day 2 and Day 3 of treatment period 2.
  Interventions: Drug: Casopitant 150 mg; Drug: Ketoconazole; Drug: Casopitant 50 mg
- Cohort 2, Group A (Placebo Comparator): Subjects will receive placebo once daily on Day 1 to Day 3 in treatment period 1. Subjects will receive ketoconazole 400 mg once daily on Day 1 to Day 9 and oral placebo once daily on Days 4, 5 and 6 in treatment period 2. There will be a 14-day washout period between treatment periods 1 and 2.
  Interventions: Drug: Ketoconazole; Drug: Casopitant 150 mg matching placebo; Drug: Casopitant 50 mg matching placebo
- Cohort 2, Group B (Experimental): In treatment period 1, subjects will receive oral casopitant 150 mg on Day 1 and 50 mg on Days 2 and 3. In treatment period 2, they will be administered ketoconazole 400 mg once daily on Day 1 to Day 9 and oral casopitant 150 mg on Day 4 and 50 mg on Days 5 and 6. There will be a 14-day washout period between treatment periods 1 and 2.
  Interventions: Drug: Casopitant 150 mg; Drug: Ketoconazole; Drug: Casopitant 50 mg

INTERVENTIONS:
Drug: Casopitant 150 mg — Casopitant 150 mg will be available as white, film-coated tablets. Casopitant tablets will be taken with 240 milliliters (mL) of water at room temperature on an empty stomach.
  Arms: Cohort 1; Cohort 2, Group B
Drug: Ketoconazole — Ketoconazole will be available as 200 mg tablets which will be taken with 240 mL of water on an empty stomach (after a 2 hour fast on Day 4 of Treatment Period 2 and after a 1 hour fast on all other dosing days).
  Other Names: Casopitant
Drug: Casopitant 150 mg matching placebo — Casopitant 150 mg matching placebo will be available as white, film-coated tablets.
  Arms: Cohort 2, Group A
Drug: Casopitant 50 mg — Casopitant 50 mg will be available as pale orange, film-coated tablets. Casopitant tablets will be taken with 240 mL of water at room temperature on an empty stomach.
  Arms: Cohort 1; Cohort 2, Group B
Drug: Casopitant 50 mg matching placebo — Casopitant 50 mg matching placebo will be available as pale orange, film-coated tablets.
  Arms: Cohort 2, Group A

SUMMARY:
Casopitant may affect liver enzymes that metabolize ketoconazole. This study is designed to test the safety and the extent of the Casopitant affect on ketoconazole levels in healthy human subjects.

ELIGIBILITY:
Inclusion criteria:

* A female subject who is non-childbearing potential or using acceptable contraceptive methods.
* Adequate organ system functions.
* Able to swallow and retain oral medication.
* Subject is able to understand and comply with protocol requirements and instruction and is likely to complete the study.

Exclusion Criteria:

* Current clinically relevant abnormality, medical condition, or circumstance that makes the subject unsuitable for the study per the study doctor.
* History of drug or other allergy which, in the opinion of the study doctor, contraindicates participation.
* Use of an investigational drug within 28 days or 5 half-lives.
* Use of prescription or non-prescription drugs, supplements or vitamins (excluding multivitamins) within 14 days, or 5 half-lives prior to first dose of study medication.
* Blood donation in excess of 500mL within 56 days prior to dosing or intends to donate within 30 days of the post-treatment follow-up visit.
* Iron deficiency.
* Positive stool for occult blood.
* Female subject who is pregnant or lactating.
* Male subject who has a history of hypogonadism.
* Positive urine drug screen.
* Positive for HIV antibody, hepatitis C antibody or hepatitis B surface antigen.
* Use of tobacco-containing products within the past 12 months prior to screening.
* History of drug or alcohol abuse or dependence within 6 months of screening.
* History or presence of uncontrolled emesis.
* Presence of active infection.
* History of cholecystectomy or biliary tract disease.
* Active peptic ulcer disease (PUD) or a history of PUD of unknown etiology.
* Any degree of heart failure.
* Consumption of any food or drink containing grapefruit or grapefruit juice, apple juice, Seville oranges, kumquats, pommelos or vegetables from the mustard green family within 7 days prior to the first dose unless prior approval is received.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2007-04-16 (Actual); Primary Completion 2007-08-27 (Actual); Study Completion 2007-08-27 (Actual)

PRIMARY OUTCOMES:
Plasma levels of casopitant and ketoconazole will be checked on Day 4 to 9 in Cohort 1. | Day 4 to 9 in Cohort 1.
Plasma levels of casopitant will be checked on Day 2 to 4 of Period 1 and | Day 2 to 4 of Period 1
casopitant and ketoconazole will be checked on Day 4 to 9 of Period 2. | Day 4 to 9 of Period 2

SECONDARY OUTCOMES:
Safety is evaluated in Cohort 1 by: - Clinical Lab Tests & Physical Exam at Screen, Day -1 & Followup (FU) | at Screen, Day -1 & Followup (FU)
- Vitals Signs monitored at Screen, Day -1, 4-7 and FU | at Screen, Day -1, 4-7 and FU
- 12 lead ECGs at Screen & FU | at Screen & FU
- Adverse Events Monitoring starting at Day 1 | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Johnson BM, Adams LM, Zhang K, Gainer SD, Kirby LC, Blum RA, Apseloff G, Morrison RA, Schutz RA, Lebowitz PF. Ketoconazole and rifampin significantly affect the pharmacokinetics, but not the safety or QTc interval, of casopitant, a neurokinin-1 receptor antagonist. J Clin Pharmacol. 2010 Aug;50(8):951-9. doi: 10.1177/0091270009353761. Epub 2010 Feb 2. PMID 20124517
- See also: Results for study 109990 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/NKV109990?search=study&search_terms=109990#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: NKV109990 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKV109990 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKV109990 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKV109990 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKV109990 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKV109990 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKV109990 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register